CLINICAL TRIAL: NCT02185703
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center Clinical Investigation to Evaluate the Performance and Safety of the Chordate System When Used in the Treatment of Acute Migraine Attacks of Moderate to Severe Intensity
Brief Title: Chordate System S020 Acute Migraine Clinical Investigation
Acronym: Amici
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow recruitment rate
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM004
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Acute Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chordate System S020 in treatment mode (Experimental)
  Interventions: Device: Chordate System S020 in treatment mode
- Chordate System S020 in placebo mode (Sham Comparator)
  Interventions: Device: Chordate System S020 in placebo mode

INTERVENTIONS:
Device: Chordate System S020 in treatment mode
  Arms: Chordate System S020 in treatment mode
Device: Chordate System S020 in placebo mode
  Arms: Chordate System S020 in placebo mode

SUMMARY:
The main purpose of the study is to evaluate the impact of treatment with the Chordate System S020 (medical device) on acute migraine headache pain.

DETAILED DESCRIPTION:
One single migraine attack will be treated either with the Chordate System S020 or with Chordate System in placebo mode.

After a screening visit, up to 3 months before treatment, eligible subjects will be asked to return to the center at the onset of their next moderate to severe migraine attack. Subjects will be re-checked for eligibility, randomized and treated at the center (treatment visit). The subjects will record their response over the next 48 hours using a diary card. A follow-up visit will be scheduled 3 to 7 days after the treatment. In addition the subjects will be contacted within 24 to 48 hours after treatment initiation via a telephone contact to discuss their health including new or ongoing AEs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with migraine, with or without aura according to International Headache Society (IHS) classification (International Classification of Headache Disorders [ICHD]-III beta).
* History of 1 to 6 migraine attacks per month for at least 12 previous months.
* At least 50% of previous migraine attacks had moderate or severe pain intensity.
* History of at least 48 hours of freedom from headache between migraine attacks.
* The majority of the previous untreated migraine attacks lasted at least 8 hours.
* Migraine onset before the age of 50 years.

Exclusion Criteria:

* History (within one year prior to inclusion into this clinical investigation) of 15 or more headache days per month (i.e. headaches of any kind).
* More than 6 days per month with non-migraine headaches (within one year prior to inclusion into this clinical investigation).
* Unable to distinguish between migraine headaches and other headache types at the onset of a migraine attack.
* Treatment with Botox in the head/neck area within 6 months of the screening visit, or between the screening and treatment visit.
* Previously treated with an implantable stimulator or any implantable devices in the head and/or neck.
* Pronounced anterior septal nasal deviation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Headache relief | 2 hours after treatment initiation
  Percentage of subjects with a decrease in migraine headache pain from severe or moderate prior treatment to mild or none at 2 hours after treatment initiation with no use of rescue medication during this time period.

SECONDARY OUTCOMES:
Pain-free rate | 2 hours after treatment initiation
  Percentage of subjects pain-free (pain intensity rated 'No pain') at 2 hours after treatment initiation with no use of rescue medication.
Incidence of recurrence | 48 hours after treatment initiation
24 hour sustained pain-free rate | 24 hours after treatment initiation
  percentage of subjects remaining pain-free
48 hour sustained pain-free rate | 48 hours after treatment initiation
  percentage of subjects remaining pain-free
Time to meaningful relief | 4 hours post-treatment initiation
Change in nausea, photophobia, phonophobia, vomiting and disability | 2 hours post-treatment initiation
Subject global impression | 48 hours post-treatment initiation.
Use of rescue medication | 48 hours post-treatment initiation
Frequency, severity, device-relationship and outcome of all adverse events | 48 hours post-treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Diener, Prof. Dr., Principal Investigator — Universitätsklinikum Essen
Locations (9):
- Germany (9):
  - Universitätsklinikum Tübingen / Zentrum für Neurologie, Tübingen, Baden-Wurttemberg
  - Praxis für Neurologie und Psychiatrie, Psychotherapie, Schmerztherapie, Erding, Bavaria
  - Neurologie- & Kopfschmerzzentrum, München, Bavaria
  - Klinikum Großhadern / Neurologische Klinik der Universität München, München, Bavaria
  - Universitätsklinikum Eppendorf, Hamburg, Hamburg
  - Migräne-Klinik Königstein, Königstein im Taunus, Hesse
  - Universitätsklinikum Essen / Neurologische Klinik, Essen, North Rhine-Westphalia
  - Praxis für spezielle Schmerztherapie, Wegberg, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin / Campus Mitte Klinik für Neurologie, Berlin, State of Berlin